CLINICAL TRIAL: NCT06317077
Title: Investigation of the Accordance Between Event Detection of prismaLINE Devices and Polysomnography Using Full Face Masks
Acronym: EventLAB FF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Löwenstein Medical Technology GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I5-R1-C-FA
Record Dates: First submitted 2024-03-02; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Sleep Apnea Syndromes
Keywords: sleep-related breathing disorders; obstructive sleep apnea; event classification; device; full face mask; apnea-hypopnea-index; polysomnography; accuracy
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Other): All participants of the clinical investigation undergo the standard stages of the clinical routine within an initial PAP therapy setting: a diagnostic night followed by a titration night (or if necessary two titration nights) with prescribed titration scheme. All participants use a full face mask of Löwenstein Medical.
  Interventions: Other: PAP therapy setting; Other: exclusive use of Löwenstein Medical full face masks

INTERVENTIONS:
Other: PAP therapy setting — Subtherapeutic phases during titration to provoke breathing events after reaching the pressure level with which the breathing events are sufficiently treated
Other: exclusive use of Löwenstein Medical full face masks — Use of a Löwenstein Medical full face mask as a requirement for participation in the clinical investigation

SUMMARY:
Sleep-related breathing disorders are highly prevalent and are usually treated with positive airway pressure (PAP) therapy. To determine the quality of therapy, PAP therapy devices measure the frequency of residual breathing events. For this purpose, breathing events of different classes are detected, counted and identified.

This clinical investigation aims to evaluate the performance of prismaLINE devices based on the accuracy of the apnea-hypopnea index (AHI) recorded in the devices. During the PAP titration night, the AHI is similarly detected via polysomnography (PSG) device and a subsequent manual scoring of the recorded PSG data. The validation of the device AHI accuracy refers to the alignment with the manually scored AHI.

Further goals of this clinical investigation are the confirmation of safety of the prismaLINE devices, the confirmation of performance and safety of LM full face masks (full face masks of the manufacturer Löwenstein Medical Technology), as well as the investigation of the influence of LM full face masks on therapy quality.

The most relevant inclusion criteria are diagnosis of a sleep-related breathing disorder and indication for therapy with continuous positive airway pressure (CPAP). Treatment takes place with prismaLINE PAP therapy devices in combination with LM full face masks.

DETAILED DESCRIPTION:
The duration of the clinical investigation per participant is two or three nights: diagnosis night with the following CPAP titration night. A further titration night (CPAP or APAP) might be necessary to find optimal therapy settings. But only the CPAP titration night with the best therapy result will be analysed.

The titration night is performed according to a predefined titration scheme. Therapy pressure will be gradually increased until breathing events are treated sufficiently. Due to the need of a certain number of remaining breathing events for sufficient performance evaluation, therapy pressure will be gradually reduced after reaching the ideal pressure level to provoke additional breathing events. The titration night is additionally monitored and recorded via polysomnography (PSG). No significant negative impact on patients' condition based on subtherapeutic phase is expected.

After the end of the clinical investigation participants will be treated according to clinical routine.

The performance of the prismaLINE therapy device will be evaluated by the accuracy of the alignment between the device AHI and the manually scored PSG AHI (using AASM hypopnea scoring rule 1A). The alignment between device AHI versus PSG AHI will be defined for coincident titration night recordings of both, therapy and PSG device.

The accuracy of the device AHI is defined by the absolute or relative deviation from the manually scored PSG AHI (ΔAHI_rel or ΔAHI_abs) and classified in acceptable, good, very good or unacceptable. The maximum deviation (ΔAHI_rel or ΔAHI_abs) is used throughout to determine the corresponding device AHI values for each category.

To achieve the primary endpoint, the proportion of the investigation population with an at least acceptable device AHI must be ≥ 80%.

ELIGIBILITY:
Inclusion Criteria:

* Polysomnographic diagnosis performed at the investigator site
* Indication for CPAP therapy (initial setting)
* Age of the participants: ≥ 18 ≤ 80 years
* AHI diagnosis night ≥ 15/h
* Capacity to consent
* Agreement to use a full face mask of Löwenstein Medical during the titration night
* Existence of a signed informed consent form for participation in the clinical investigation and a signed declaration of consent for the use of data within the scope of the DSGVO

Exclusion Criteria:

* Presence of a contraindication to CPAP therapy
* Participation in another clinical investigation that influences the adjustment to CPAP therapy by stipulate device settings or titration
* pregnant or breastfeeding woman

Inclusion Criteria Statistical Evaluation:

* AHI PSG (diagnosis and therapy) and AHI of the device (therapy) are completely available
* Evaluation of the mask/device functionalities is available
* Clear documentation of (predictable) adverse events and (predictable) adverse device effects
* Existence of a signed informed consent form for participation in the clinical investigation and a signed declaration of consent for the use of data within the scope of the DSGVO
* Reliable evaluation of the polysomnography (titration night) is possible: no missing signals, good signal quality, no deviation of the applied CPAP pressure course from the course specified for the clinical investigation
* Total sleep time during the titration night ≥ 4 hrs
* Proportion of the therapy time with high leakage (more than 50 l/min) < 10%
* The quality assurance process did not identify any deviations from the source data that could not be corrected

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Delta AHI [n/h]= Difference of device AHI (prismaLINE devices of the type WM100TD) and the manual scored AHI of polysomnographic data identified in the Matlab-based SOMNOmat tool | 1 night
  comparison of PSG AHI (according to AASM hypopnea scoring rule 1A and 1B) and device AHI for the period in which the records of both devices are available

SECONDARY OUTCOMES:
N_AE device [n]= number and severity of occurred (predictable) adverse events and (predictable) adverse device effects, counted during study duration | 1 night
  Confirmation of safety of the prisma therapy devices (type WM100TD)
Mask fit score= Leakage, pressure points, stable pressure level, comfort determined via questionnaire | 1 night
  Confirmation of performance of the full face masks of Löwenstein Medical
N_AE mask [n]= number and severity of occurred (predictable) adverse events and (predictable) adverse device effects, counted during study duration | 1 night
  Confirmation of safety of the full face masks of Löwenstein Medical
Delta AI [n/h]= difference of apnea-indices (obstructive/central/mixed) between the therapy device and the manually evaluated PSG data identified in the Matlab-based tool SOMNOmat | 1 night
  Investigation of the accordance of the individual event indices of the synchronized device and PSG files
Delta HI [n/h]= difference of hypopnea-indices (obstructive/central) between the therapy device and the manually evaluated PSG data identified in the Matlab-based tool SOMNOmat | 1 night
  Investigation of the accordance of the individual event indices of the synchronized device and PSG files
Delta Event_individual [n]= difference of the number (with time, duration, type) of residual breathing events (apneas/hypopneas) device vs. PSG identified in the Matlab-based tool SOMNOmat | 1 night
  Comparison of all AHI-relevant individual events of the synchronized device and PSG files
N_influenced phases [n]= number (with time, duration, type) of phases with significant deviations between the synchronized device and PSG files identified in the Matlab-based tool SOMNOmat | 1 night
  investigation of influencing factors for accordance between therapy device and the polysomnography (e.g. phases with increased pressure or increased leakage)
Delta AHI_1A [n/h]= difference between apnea indices using scoring rule 1A from AASM manual version 3.0 | 1 night
  investigation of impact of AASM hypopnea scoring rules 1A from AASM manual, version 3.0
Delta AHI_1B [n/h]= difference between apnea indices using scoring rule 1B from AASM manual version 3.0 | 1 night
  investigation of impact of AASM hypopnea scoring rules 1B from AASM manual, version 3.0
Delta AHI_mean [n/h]= difference between apnea indices using mean of scoring rule 1A and 1B from AASM manual version 3.0 (AHI_1A + AHI_1B)/2 | 1 night
  investigation of impact of AASM hypopnea mean of scoring rule 1A and 1B from AASM manual, version 3.0
Delta AHI_Routine [n/h]= difference between unmachined apnea indices of device and PSG | 1 night
  comparison of original device AHI and PSG AHI to investigate the alignment of routine device AHI with routine PSG AHI (1A/1B)
N_impact factors [n]= number and type of factors that can increase the risk for sleep related breathing disorders like comorbidities and smoking | 1 night
  investigation of influencing factors and identification of confounders
corr_flow-sleep= correlation between flow signal and sleep state | 1 night
  identification of correlation between flow signal and sleep state
corr_marker= correlation between diagnostic sleep apnea syndrom markers with medical history data, biomarkers of the diagnostic night, therapy pressure and sleep stage | 1 night
  identification of correlation of modern versus classic diagnostic sleep apnea syndrom markers

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Randerath, Prof. Dr., Principal Investigator — Krankenhaus Bethanien (Solingen), Klinik für Pneumologie und Allergologie/Zentrum für Schlaf- und Beatmungsmedizin
Locations (1):
- Krankenhaus Bethanien, Solingen, North Rhine-Westphalia, Germany